CLINICAL TRIAL: NCT04905797
Title: Aspects of Self-harm - Cognition, Imaging and Treatability
Status: Recruiting | Type: Observational
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other)
Responsible Party: Principal Investigator, Sofie Westling, MD, associate professor, Region Skane
Other Study IDs: 2020-02732
Record Dates: First submitted 2021-04-29; First posted 2021-05-28 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Self-Harm, Deliberate; Non-Suicidal Self Injury; Attempt Suicide; Personality Disorders
MeSH Terms: conditions — Self-Injurious Behavior; Suicide, Attempted; Personality Disorders | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Deliberate self-harm: Individuals with psychiatric disorders and persistent DSH
  Interventions: Diagnostic Test: Emotional Stop Signal Task; Diagnostic Test: Magnetic Resonance Imaging; Other: World Health Organizations Disability Assessment Schedule (WHODAS 2.0); Diagnostic Test: Personality Inventory for DSM-5 (PID-5); Diagnostic Test: Stop Signal Task (CANTAB); Diagnostic Test: Intra-Extra Dimensional Set Shift (CANTAB); Diagnostic Test: Spatial Working Memory Test (CANTAB); Diagnostic Test: Multitasking Test (CANTAB); Diagnostic Test: Cambridge Gambling Task Test
- Clinical cases who ceased self-harm: Individuals with psychiatric disorders who have ceased DSH
  Interventions: Diagnostic Test: Emotional Stop Signal Task; Diagnostic Test: Magnetic Resonance Imaging; Other: World Health Organizations Disability Assessment Schedule (WHODAS 2.0); Diagnostic Test: Personality Inventory for DSM-5 (PID-5); Diagnostic Test: Stop Signal Task (CANTAB); Diagnostic Test: Intra-Extra Dimensional Set Shift (CANTAB); Diagnostic Test: Spatial Working Memory Test (CANTAB); Diagnostic Test: Multitasking Test (CANTAB); Diagnostic Test: Cambridge Gambling Task Test
- Clinical cases with no self-harm: Individuals with psychiatric disorders who never had DSH
  Interventions: Diagnostic Test: Emotional Stop Signal Task; Diagnostic Test: Magnetic Resonance Imaging; Other: World Health Organizations Disability Assessment Schedule (WHODAS 2.0); Diagnostic Test: Personality Inventory for DSM-5 (PID-5); Diagnostic Test: Stop Signal Task (CANTAB); Diagnostic Test: Intra-Extra Dimensional Set Shift (CANTAB); Diagnostic Test: Spatial Working Memory Test (CANTAB); Diagnostic Test: Multitasking Test (CANTAB); Diagnostic Test: Cambridge Gambling Task Test
- Healthy controls: Healthy controls who never had DSH
  Interventions: Diagnostic Test: Emotional Stop Signal Task; Diagnostic Test: Magnetic Resonance Imaging; Other: World Health Organizations Disability Assessment Schedule (WHODAS 2.0); Diagnostic Test: Personality Inventory for DSM-5 (PID-5); Diagnostic Test: Stop Signal Task (CANTAB); Diagnostic Test: Intra-Extra Dimensional Set Shift (CANTAB); Diagnostic Test: Spatial Working Memory Test (CANTAB); Diagnostic Test: Multitasking Test (CANTAB); Diagnostic Test: Cambridge Gambling Task Test

INTERVENTIONS:
Diagnostic Test: Emotional Stop Signal Task — Emotional Stop Signal Task (modified version from CANTAB). Outcome Measure is commission and omission errors - higher score (percentage) indicate worse performance.
Diagnostic Test: Magnetic Resonance Imaging — Functional Magnetic Resonance Imaging (fMRI) Diffusion Tensor Imaging (DTI) Volumetry
Other: World Health Organizations Disability Assessment Schedule (WHODAS 2.0) — Self-reported data on World Health Organizations Disability Assessment Schedule - 36 items self-administered (WHODAS 2.0). Assessing six domains of functional disability in daily life. Each item is rated on a Likert scale ranging from 0-4. Total range 0 - 144. High scores scores indicate more severe disability.
Diagnostic Test: Personality Inventory for DSM-5 (PID-5) — Self-rated personality traits through Personality Inventory for DSM-5 (PID-5). Self-reported scores on domains of personality traits. Higher scores in one domain indicate more pronounced traits in this domain.
Diagnostic Test: Stop Signal Task (CANTAB) — The estimate of time where an individual can successfully inhibit their responses 50% of the time.
Diagnostic Test: Intra-Extra Dimensional Set Shift (CANTAB) — 1. The number of trials for which the outcome was an incorrect response (subject pressed the incorrect button within the response window), calculated across all assessed trials.
  2. The total number of times that the subject chose a wrong stimulus - i.e. one incompatible with the current rule, adjustment for every stage that was not reached.
Diagnostic Test: Spatial Working Memory Test (CANTAB) — 1. The number of times the subject incorrectly revisits a box in which a token has previously been found. Calculated across all assessed four, six and eight token trials.
  2. The number of times a subject begins a new search pattem from the same box they started with previously. If they always begin a search from the same starting point, we infer that the subject is employing a planned strategy for finding the tokens. Therefore, a low score indicates high strategy use (1 = they always begin the search from the same box), a high score indicates that they are beginning their searches from many different boxes. Calculated across assessed trials with 6 tokens or more.
Diagnostic Test: Multitasking Test (CANTAB) — 1. The number of trials for which the outcome was an incorrect response.
  2. The median latency of response (from stimulus appearance to button press). Calculated across all correct, assessed trials.
  3. The difference between the median latency of response on the trials that were congruent versus the trials that were incongruent. A positive score indicates that the subject is faster on congruent trials and a negative score indicates that the subject is faster on incongruent trials. A higher incongruency cost indicates that the subjects take longer to process conflicting information.
  4. The difference between the median latency of response during assessed blocks in which both rules are used versus assessed blocks in which only a single rule is used. A positive score indicates that the subject responds more slowly during multitasking blocks and indicates a higher cost of managing multiple sources of information.
Diagnostic Test: Cambridge Gambling Task Test — 1. The proportion (0 - 1) of all trials where the subject chose the majority box color. Calculated over all assessed trials from both the ascending and descending conditions in which the number of boxes of each color differed.
  2. Risk adjustment is a measure of sensitivity to risk, based on the ability to modify choices in the light of information about the probability of different outcomes and to track the optimal outcome on eaeh trial. The measure is calculated from the average proportion of points that the subject ehose to bet with, taking into aeeount the number of colored boxes in the majority.
  3. Allows for the dissociation between risk taking and impulsivity by determining whether subjects simply just place a bet at the first opportunity. Calculated as CGT Risk Taking for all trials from the descending condition minus CGT Risk Taking for all trials from the ascending condition.

SUMMARY:
Deliberate self-harm (DSH) is a common symptom in psychiatric disorders. This study aim at increased understanding of parameters associated with DSH with the long term goal to potentially improve and possibly personalise its treatment.

In short, the study will characterise cognitive, psychiatric and demographic factors with focus on executive function and will compare results from individuals with DSH, individuals who have ceased DSH as well as psychiatric patients without DSH and individuals who never engaged in DSH. Adequate statistical tests will be used to compare groups.

Participants will be interviewed by a trained physician for basic medical history, history of self-harm and treatment for that, demographic data and diagnostic evaluation. Thereafter the participants will undergo standardised neuropsychological testing focusing on emotional response inhibition, decision making and risk taking, attention set shifting, working memory, inhibition and planning. Some participants will redo parts of this testing during fMRI, as well as undergo DTI and volumetry.

DETAILED DESCRIPTION:
Deliberate self-harm (DSH) is a common symptom in psychiatric disorders. Today, there is not sufficient knowledge as to why an individual continues to suffer from DSH, DSH is reduced or even ceased - regardless given treatment or not. The overall aim of this project is to characterise cognitive, psychiatric and demographic factors as well as perform brain imaging in individuals currently suffering from DSH, individuals with a prior history of DSH, individuals with psychiatric disease but no DSH and healthy individuals. The intention is to gain more knowledge on factors associated with DSH and thereby potentially improve and possibly personalize treatment.

The following hypotheses will be tested:

Individuals currently suffering from DSH have lower scores on executive function than individuals with a prior history of DSH, individuals with psychiatric disease but no DSH and healthy individuals.

Individuals currently suffering from DSH have lower level daily life functioning and more severe psychiatric symptoms than individuals with a prior history of DSH, individuals with psychiatric disease but no DSH and healthy individuals.

Individuals currently suffering from DSH have higher scores of negative affectivity, lower scores of antagonism and lower scores of disinhibition measured with Personality Inventory for DSM-5 than individuals with a prior history of DSH, individuals with psychiatric disease but no DSH and healthy individuals.

Individuals currently suffering from DSH have, when executing the neurocognitive tests in hypothesis 1, a significant lower blood flow in the prefrontal network, than individuals with a prior history of DSH, individuals with psychiatric disease but no DSH and healthy individuals.

Individuals currently suffering from DSH have a decrease in local cerebral white matter compared to individuals with a prior history of DSH, individuals with psychiatric disease but no DSH and healthy individuals.

Material:

The aim is to recruit 300 participants in total, 75 participants to each group:

1. individuals with psychiatric disorders and persistent DSH
2. individuals with psychiatric disorders who have ceased DSH
3. individuals with psychiatric disorders who never had DSH
4. healthy controls who never had DSH

Participants will be interviewed by a trained physician for basic medical history, history of self-harm and treatment for that, demographic data and diagnostic evaluation. Thereafter the participants will undergo standardised neuropsychological testing focusing on emotional response inhibition, decision making and risk taking, attention set shifting, working memory, inhibition and planning. Some participants will redo parts of this testing during fMRI, as well as undergo DTI and volumetry.

ELIGIBILITY:
Inclusion criteria for persistent DSH group:

* Adults 18-65 years.
* Ability to leave informed consent.
* Understands and uses the Swedish language without significant difficulties.
* Psychiatric disorder and ongoing treatment at an adult psychiatric clinic.
* DSH at least five times during the last three months, and DSH at least ten times during at least one year.

Exclusion criteria for persistent DSH group:

* No history of DSH, and/or DSH fewer than five times during the last three months and fewer than ten times during at least one year
* Diagnosis of Intellectual disability
* Diagnosis of chronic psychotic disorder
* Hearing disability, visual impairment or motor disorder that rules out the ability to complete neurocognitive tasks

Inclusion criteria for those who have ceased DSH group:

* Adults 18-65 years.
* Ability to leave informed consent.
* Understands and uses the Swedish language without significant difficulties.
* Psychiatric disorder and ongoing treatment at an adult psychiatric clinic.
* No DSH during the last three months, but DSH at least ten times during at least one year.

Exclusion criteria for those who have ceased DSH group:

* Any DSH during the last three months, and/or fewer than ten times during the at least one year
* Diagnosis of Intellectual disability
* Diagnosis of chronic psychotic disorder
* Hearing disability, visual impairment or motor disorder that rules out the ability to complete neurocognitive tasks

Inclusion criteria for psychiatric disorder with no history of DSH group:

* Adults 18-65 years.
* Ability to leave informed consent.
* Understands and uses the Swedish language without significant difficulties.
* Psychiatric disorder and ongoing treatment at an adult psychiatric clinic.

Exclusion criteria for psychiatric disorder with no history of DSH group:

* Any DSH during the last three months, and more than two times during lifetime
* Diagnosis of Intellectual disability
* Diagnosis of chronic psychotic disorder
* Hearing disability, visual impairment or motor disorder that rules out the ability to complete neurocognitive tasks

Inclusion criteria for healthy control group:

* Adults 18-65 years.
* Ability to leave informed consent.
* Understands and uses the Swedish language without significant difficulties.

Exclusion criteria for healthy control group:

* Diagnosed with any psychiatric disorder
* Any DSH during the last three months, and more than two times during lifetime
* Hearing disability, visual impairment or motor disorder that rules out the ability to complete neurocognitive tasks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Clinical participants will be recruited though a cohort listed on an out-patient psychiatric clinic in Lund.
  Healthy controls will be recruited through through fliers placed on public advertisement boards.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-04-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Executive functioning | Up to 1 hour
  Scores on cognitive tests measuring executive functioning
Level of function in daily life | 30 days
  Scores on WHODAS 2.0
Personality traits | More than 1 year (stable)
  Scores on Personality Inventory for DSM-5
Blood flow | Up to 1 hour
  Blood flow in prefrontal cortex during neurocognitive tests
Volumetry | Up to 1 hour
  Volumes of local cerebral white matter

CONTACTS AND LOCATIONS:
Overall Officials: Sofie Westling, MD PhD, Principal Investigator — Region Skåne
Locations (1):
- Psykiatri och habilitering, Region Skåne, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Data not protected by Swedish law of patient secrecy can be shared after analyses has been completed and man scripts accepted for publication

REFERENCES:
- [Background] Allen KJ, Hooley JM. Inhibitory control in people who self-injure: evidence for impairment and enhancement. Psychiatry Res. 2015 Feb 28;225(3):631-7. doi: 10.1016/j.psychres.2014.11.033. Epub 2014 Dec 2. PMID 25510907
- [Background] Allen KJ, Hooley JM. Negative mood and interference control in nonsuicidal self-injury. Compr Psychiatry. 2017 Feb;73:35-42. doi: 10.1016/j.comppsych.2016.10.011. Epub 2016 Nov 4. PMID 27888700
- [Background] Allen KJD, Hooley JM. Negative Emotional Action Termination (NEAT): Support for a Cognitive Mechanism Underlying Negative Urgency in Nonsuicidal Self-Injury. Behav Ther. 2019 Sep;50(5):924-937. doi: 10.1016/j.beth.2019.02.001. Epub 2019 Feb 14. PMID 31422848
- [Background] McHugh CM, Chun Lee RS, Hermens DF, Corderoy A, Large M, Hickie IB. Impulsivity in the self-harm and suicidal behavior of young people: A systematic review and meta-analysis. J Psychiatr Res. 2019 Sep;116:51-60. doi: 10.1016/j.jpsychires.2019.05.012. Epub 2019 May 17. PMID 31195164
- [Background] Ackerman JP, McBee-Strayer SM, Mendoza K, Stevens J, Sheftall AH, Campo JV, Bridge JA. Risk-sensitive decision-making deficit in adolescent suicide attempters. J Child Adolesc Psychopharmacol. 2015 Mar;25(2):109-13. doi: 10.1089/cap.2014.0041. Epub 2014 Sep 29. PMID 25265242
- [Background] Oldershaw A, Grima E, Jollant F, Richards C, Simic M, Taylor L, Schmidt U. Decision making and problem solving in adolescents who deliberately self-harm. Psychol Med. 2009 Jan;39(1):95-104. doi: 10.1017/S0033291708003693. Epub 2008 Jun 23. PMID 18570698
- [Background] Chamberlain SR, Odlaug BL, Schreiber LR, Grant JE. Clinical and neurocognitive markers of suicidality in young adults. J Psychiatr Res. 2013 May;47(5):586-91. doi: 10.1016/j.jpsychires.2012.12.016. Epub 2013 Jan 26. PMID 23357208
- [Background] Fikke LT, Melinder A, Landro NI. Executive functions are impaired in adolescents engaging in non-suicidal self-injury. Psychol Med. 2011 Mar;41(3):601-10. doi: 10.1017/S0033291710001030. Epub 2010 May 19. PMID 20482935
- [Background] Gvirts HZ, Braw Y, Harari H, Lozin M, Bloch Y, Fefer K, Levkovitz Y. Executive dysfunction in bipolar disorder and borderline personality disorder. Eur Psychiatry. 2015 Nov;30(8):959-64. doi: 10.1016/j.eurpsy.2014.12.009. Epub 2015 Oct 21. PMID 26647872
- [Background] Thompson C, Ong ELC. The Association Between Suicidal Behavior, Attentional Control, and Frontal Asymmetry. Front Psychiatry. 2018 Mar 14;9:79. doi: 10.3389/fpsyt.2018.00079. eCollection 2018. PMID 29593586